CLINICAL TRIAL: NCT07318142
Title: Evaluation of the Effectiveness of Vestibular Rehabilitation With Virtual Reality Systems in Individuals With Visually Induced Motion Sickness
Brief Title: Virtual Reality in the Rehabilitation of Visually Induced Motion Sickness
Acronym: VIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Rukiye Tanisir Disci, Research Assistant, Istanbul Aydın University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28/2024
Record Dates: First submitted 2025-11-21; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-01

CONDITIONS: Motion Sickness, Space; Visually Induced Motion Sickness; Vestibular Rehabilitation in MS
Keywords: Visually induced motion sickness; virtual reality; vestibular rehabilitation
MeSH Terms: conditions — Space Motion Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality-Based Vestibular Rehabilitation (Experimental): The study group consisted of individuals with visually induced motion sickness (VIMS). Participants underwent a four-week virtual reality-based rehabilitation program consisting of eight sessions (30 minutes per session). The effects of VR exposure were assessed using posturography.
  Interventions: Other: The effects of virtual reality exposure were assessed using posturography.

INTERVENTIONS:
Other: The effects of virtual reality exposure were assessed using posturography. — The study group (individuals with VIMS) underwent a four-week VR rehabilitation program consisting of 8 sessions, each lasting 30 minutes.

SUMMARY:
In recent years, rapidly advancing virtual reality (VR) technology has been widely used in many fields, from education to health and from entertainment to therapeutic applications, by creating interactive and highly immersive digital environments. However, the increasing use of VR systems has also been associated with physiological side effects. One of these is Visually Induced Motion Sickness (VIMS), a syndrome characterized by symptoms such as eye strain, fatigue, dizziness, headache, and nausea, especially when individuals experience a sense of motion in virtual environments despite physical immobility. VIMS is thought to occur due to sensory conflicts among the visual, vestibular, and motor systems, and its severity may vary depending on individual factors and the intensity of the visual motion cues.

The aim of this study is to evaluate the effect of a VR-based vestibular rehabilitation program on symptoms associated with VIMS. The VR stimuli consist of real travel videos available on the YouTube VR platform. To enhance familiarity and the sense of presence, 360° videos depicting scenes from Istanbul, Turkey were selected and categorized based on difficulty level.

The study includes two groups: a control group of healthy individuals and an experimental group of individuals diagnosed with VIMS. All participants undergo baseline assessments. The experimental group receives a VR-based vestibular rehabilitation program for 4 weeks, delivered twice per week, with each session lasting 30 minutes. The intervention uses a VR headset and consists of progressively challenging visual motion stimuli.

The effectiveness of the intervention will be evaluated using both subjective and objective outcome measures, including the Simulator Sickness Questionnaire (SSQ), visual analog scale (VAS) symptom ratings, and static posturography assessments (Balance Screening and Limits of Stability - Reaction Time). Pre- and post-intervention assessments will be compared within and between groups to determine the impact of the rehabilitation program.

This study is designed to contribute to the understanding of VR-based vestibular rehabilitation approaches and to support the development of safer and more effective VR applications.

DETAILED DESCRIPTION:
This prospective single-arm interventional study was designed to evaluate the effects of a virtual reality (VR)-based rehabilitation program in individuals with visually induced motion sickness (VIMS). Following baseline assessment, participants underwent a structured VR rehabilitation protocol over a four-week period.

The intervention consisted of eight supervised sessions, conducted twice weekly, with each session lasting approximately 30 minutes. VR exposure was delivered using a head-mounted display and included visually complex motion stimuli aimed at gradually increasing visual-vestibular tolerance. The difficulty and visual motion intensity were progressed based on participant tolerance throughout the program.

Outcome assessments were performed at baseline and after completion of the intervention period. Postural control was objectively evaluated using static posturography, and symptom severity was monitored using validated subjective assessment tools.

This design allowed for within-subject comparison of pre- and post-intervention outcomes to examine the potential effectiveness of VR-based rehabilitation in reducing VIMS-related symptoms and improving postural stability.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria (n = 46)

* Aged between 18 and 30 years
* No history of otologic surgery
* No history of orthopedic surgery related to the lower extremities
* No claustrophobia
* Female participants not in menstrual or premenstrual periods
* No diagnosed neurological disorders/diseases (e.g., MS, epilepsy, cerebrovascular accident, etc.)
* No diagnosed peripheral vestibular pathologies such as Meniere's disease, BPPV, or vestibular neuritis (participants' lack of peripheral vestibular pathology confirmed by audiovestibular vHIT testing)
* No spontaneous nystagmus

Study Group (21.8 ± 2.9 years, n = 23) Inclusion Criteria

VIMSSQ Questionnaire:

Participants answered "occasionally" or "frequently" to Question 2

Control Group (23.7 ± 3.3 years, n = 23) Inclusion Criteria

GUHHYSA Questionnaire:

Participants answered "never" to Question 2

Exclusion Criteria:

* History of otologic surgery
* History of orthopedic surgery in the lower extremities
* Presence of claustrophobia
* Female participants in menstrual or premenstrual periods
* Diagnosed neurological disorders/diseases (e.g., MS, epilepsy, cerebrovascular accident, etc.)
* Diagnosed peripheral vestibular pathologies such as Meniere's disease, BPPV, or vestibular neuritis (as confirmed by audiovestibular vHIT testing)
* Presence of spontaneous nystagmus
* Participants who did not sign the informed consent form

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Simulator Sickness Questionnaire (SSQ) Total Score Unit of Measure: points (0-42; higher scores indicate worse symptoms) Time Frame: Baseline and 4 weeks | Time Frame: Baseline and 4 weeks
  Assessment of VIMS-related symptoms using the Simulator Sickness Questionnaire.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Symptom Score | Time Frame: Baseline and 4 weeks
  Self-reported symptom severity using a 0-10 point Visual Analog Scale. Unit of Measure: points (0 = no symptoms, 10 = worst symptoms; higher scores indicate worse symptoms)

OTHER OUTCOMES:
Static Posturography - Balance Screening Score | Time Frame: Baseline and 4 weeks
  Postural stability is objectively assessed using static posturography balance screening parameters. The balance screening score is expressed in degrees and is calculated based on individual anthropometric characteristics, including body height and weight. Higher scores indicate poorer postural stability.
Static Posturography - Limits of Stability Reaction Time | Time Frame: Baseline and 4 weeks
  Assessment of reaction time during limits of stability testing. Unit of Measure: seconds (lower values indicate better performance)

CONTACTS AND LOCATIONS:
Overall Officials: Rukiye Tanisir Disci, Principal Investigator — Istanbul Aydın University
Locations (1):
- Istanbul Aydin University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data that underlie the results of this study, including baseline characteristics, Simulator Sickness Questionnaire scores, static posturography parameters (Balance Screening and Limit of Stability - Reaction Time), and VAS symptom ratings.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available beginning 6 months after publication of the main results and will remain accessible for 5 years.
Access Criteria: Data will be available upon reasonable request to the corresponding author (Dr. Audiologist Rukiye Tanisir Disci, Istanbul Aydın University) via institutional email, after signing a data access agreement ensuring participant confidentiality.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT07318142/Prot_SAP_ICF_000.pdf